CLINICAL TRIAL: NCT04089670
Title: Online Acceptance and Commitment Therapy for Chronic Pain in Sample of People With Chiari Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Utah State University (Other); Conquer Chiari (Unknown)
Responsible Party: Principal Investigator, Douglas L. Delahanty, Professor and Associate Vice President of Research, Kent State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-171
Record Dates: First submitted 2019-05-09; First posted 2019-09-13 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain; Chiari Malformation
Keywords: Chronic Pain; Acceptance and Commitment Therapy; Sleep Dysfunction; Online Intervention
MeSH Terms: conditions — Chronic Pain; Arnold-Chiari Malformation; Parasomnias

STUDY DESIGN:
Intervention Model Description: Two groups are created through randomization to either the treatment group or the control group. The treatment includes 8 online intervention modules that are administered weekly for 8 weeks. A 7-day sleep diary is administered one week prior to the intervention and one week after the intervention. The control group completes the online sleep diaries and all the same assessments as the treatment group. At the end of the 1 month follow-up they are given the opportunity to receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Acceptance and Commitment Therapy Intervention (Active Comparator): This online Acceptance and Commitment Therapy intervention is delivered over 8 weeks, in 8 15-minute modules. Each module has a practice assignment at the end with the goal of having the participant engage in the material over the next week. Additionally, each participant will receive a weekly call for the duration of the intervention (i.e., 9 phone calls, one introduction phone call, 8 module related phone calls) from a Master's-level clinical student who will serve as the participants "phone coach." During the call the clinical student will be able to help troubleshoot any technical difficulties being experienced, as well as clarify any questions about the material being taught in the intervention.
  Interventions: Behavioral: Online Acceptance and Commitment Therapy Intervention
- Control (No Intervention): Participants in this arm of the study will complete the same sleep diaries and questionnaires at the same time points as the intervention group, but will not be administered the intervention modules and will not receive any phone coaching. When they have completed the 1-month follow-up they will be offered the intervention.

INTERVENTIONS:
Behavioral: Online Acceptance and Commitment Therapy Intervention — The intervention includes 8 modules (i.e, Away Moves, Letting Go of Control, Noticing Hooks, Stepping Back, Your Values, How You Want to Act, Goal Setting, and Making Commitments). "Away Moves" and "Letting Go of Control," helps establish creative hopelessness, where one abandons futile struggles against negative internal experiences and accepts new solutions. These two modules also help identify experiential avoidance and focus on acceptance. "Noticing Hooks" and "Stepping Back" focus on defusion, self as context, and mindfulness. While, mindfulness is overtly addressed in the module "Stepping Back" it is weaved through each module. "Your Values" and "How You Want to Act" focus on helping participants identify their values. "Goal Setting" and "Making Commitments" focus on committed action. Each module ends with a practice assignment which participants are asked to engage in over the next week.
  Arms: Online Acceptance and Commitment Therapy Intervention

SUMMARY:
Twenty percent of US adults report chronic pain symptoms. Both psychological symptoms and sleep issues commonly co-occur with chronic pain. Chronic pain is a frequently reported symptoms of Chiari Malformation (CM); however, the cause of pain symptoms is not fully understood, and pain is not associated with the extent of neural abnormality in CM.

ACT is not a set of techniques, but rather a way of thinking. ACT encourages acceptance, as opposed to avoidance of unwanted feelings, all in the context of mindfulness (i.e., being aware of one's present environment and in tune with internal thoughts and emotions). ACT has been found to be successful at reducing pain perceptions and targeting multiple symptoms at one time. However, ACT has not been examined in CM and it is unknown whether ACT will improve sleep as well as pain-related symptoms. The purpose of the current study is to assess the efficacy of an online ACT intervention at reducing pain interference and sleep dysfunction symptoms in a sample with CM. It is hypothesized that CM patients may benefit from Acceptance and Commitment Therapy (ACT). More specifically it is hypothesized that the treatment group will report significantly less pain interference and psychological flexibility compared to the control group. It is also hypothesize that ACT will mediate the relationship between sleep dysfunction and pain interference.

Based on power analyses the sample size will be 56. The sample will be recruited online and randomized to the treatment or control group. The intervention will consist of eight modules that are administered weekly over eight weeks. Additionally, a 7-day sleep diary will be administered the week prior to the intervention and the week after the intervention. Follow up assessments will be administered upon completion of the 8-week intervention (at the beginning of week 9), 1-month after, and 3 months after the completion of the intervention.

DETAILED DESCRIPTION:
Chronic pain is extremely prevalent with 20% of adults in the US reporting symptoms (Dahlhamer, 2018). Further, when accounting for lost productivity and direct health care costs, the financial burden of chronic pain has been estimated to be $560-$630 billion annually (Gaskin & Richard, 2011). A myriad of factors contribute to chronic pain including psychological symptoms and sleep. Though psychological symptoms often co-occur with chronic pain with rates estimated to be as high as 50% (Kroenke et al., 2011), chronic pain co-occurs at an even higher rate with sleep dysfunction (89%) (van Hecke, Torrance, & Smith, 2013). Sleep is believed to have a reciprocal relationship with pain, such that pain impacts sleep and sleep impacts future pain (M. T. Smith, Huang, & Manber, 2005) reciprocal relationship makes sleep an essential aspect of chronic pain that warrants attention in interventions. One intervention that has shown particular promise in treating chronic pain is Acceptance and Commitment Therapy (ACT).

ACT is not a set of techniques, but rather an orientation. This orientation focuses on living a fulfilling life by way of living in line with one's values. In addition to living a life based on values, ACT encourages acceptance, as opposed to avoidance of unwanted feelings, all in the context of mindfulness (i.e., being aware of one's present environment and in tune with internal thoughts and emotions) (S. C. Hayes, Luoma, Bond, Masuda, & Lillis, 2006). Since the focus is on an orientation rather than specific techniques, ACT can be used as a transdiagnostic intervention, targeting multiple symptoms at one time. As previously noted, chronic pain is a complex diagnosis, with many interacting factors including psychological symptoms, sleep, and decreased daily functioning. ACT effectively treats the complex presentation of chronic pain. Chronic pain already costs society billions of dollars annually and administering psychological interventions are expensive and may not be available to all those in need. Online ACT interventions remedy this issue by providing services to those where treatment may not be readily available for a fraction of the price.

Though a handful of studies have explored different online ACT interventions, and found them to be efficacious, however, they have been unable to flexibly address individual differences in symptom presentations as they present the same information regardless of the participant's symptoms (Buhrman et al., 2013; S. Hayes et al., 2014; Kristjánsdóttir et al., 2013; Lin, Klatt, McCracken, & Baumeister, 2018; Simister et al., 2018; Trompetter, Bohlmeijer, Veehof, & Schreurs, 2015). Additionally, all prior online ACT interventions for chronic pain focused on pain primarily, providing examples and metaphors around the experience of pain. The aim is to administer an intervention that broadly teaches ACT philosophies without focusing only on pain, addressing individual differences in symptom presentation and allowing for personalization. The goal is to address chronic pain but to also facilitate the generalization of skills to comorbid conditions that often perpetuate the experience of chronic pain (i.e., depression, anxiety, and sleep dysfunction). Efficacy will be assessed through reductions in pain interference as well as comorbid conditions (i.e., sleep dysfunction, anxiety and depression).

Chronic pain is a commonly reported symptom of Chiari Malformation (CM). This under-researched diagnosis is characterized by the cerebellar tonsils descending 5mm or more into the spinal canal and impacts approximately 3.25 million people or 1% of the US population (B. W. Smith et al., 2013). Although chronic pain is commonly reported in CM, the etiology of a symptomatic presentation is not fully understood, and there is no direct relationship between the extent of descension of the cerebellar tonsils and pain. Regardless of elucidating the etiology of pain in CM, those with this complex chronic pain diagnosis would likely benefit from psychological and behavioral based interventions. Further, no ACT based intervention has been administered to a sample with Chiari Malformation. The purpose of the current study is to assess the efficacy of an online broad ACT intervention on a sample with Chiari Malformation.

Aim 1: Determine the efficacy and breadth of an online ACT intervention in decreasing pain interference, sleep dysfunction, depression, and anxiety.

Hypothesis 1: The treatment group will report significantly less pain interference, sleep dysfunction, depression, and anxiety compared to the control group.

Aim 2: Assess psychological flexibility as a mechanism of ACT. Hypothesis 2: Psychological flexibility will mediate the trajectories in pain interference, sleep dysfunction, depression, and anxiety over time.

The following is a summary of the protocol:

(Part 1): (Both Treatment & Waitlist Control Groups) Consent will be established via an online form. Once consent is acquired a set of questionnaires covering demographics, as well as quality of life, pain interference, pain acceptance, anxiety, depression, stress, and sleep; taking approximately 30 - 45 minutes will be completed. Internet access is required to complete these questionnaires on a computer, tablet, or mobile phone.

(Part 2): (Both Treatment & Waitlist Control Groups) Next, a 7-day sleep diary will be completed. A Qualtrics link will be emailed out each morning (the email will be sent out by midnight the night prior) that will lead to a 2-5 minute survey (11 questions). This survey is to be completed as close to waking as possible to obtain the most accurate information. Once the final day of the sleep diary is completed, randomization into the treatment or control group will occur. The treatment will begin the following Friday after the completion of the sleep diary.

(Part 3): (Treatment Group alone) Once a week, for the next 8 weeks, a short battery of questionnaires, followed by the online intervention (taking a combined total of approximately 30-45 minutes a week) will be completed. The Qualtrics link will be sent via email every Friday morning. If the assessment and intervention has not been completed by the end of day 4 (Monday), a phone call will serve as a reminder and to answer any technical or unresolved issues. Each online intervention ends with a practice assignment for the remainder of the week. The treatment group will receive a weekly call from a Master's-level clinical student; the time of this call will be set up online during the first session in Part 3. During the call will serve to help troubleshoot any technical difficulties, as well as clarify any questions about the material being taught in the intervention.

(Waitlist Control Group) Each week for the next 8 weeks a short battery of questionnaires taking approximately 10-15 minutes will be completed. Technical issues will be remedied through communication with the the study email (chiaristudy@gmail.com).

(Part 4): (Both Treatment & Waitlist Control Groups) At the beginning of the 9th week, an immediate follow-up set questionnaires (same as in Part 1) will be administered.

(Part 5): (Both Treatment & Waitlist Control Groups) Next, a 7-day sleep diary will again be completed, taking approximately the 2-5 minutes (11 questions), and completed as close to waking as possible to provide the most accurate information.

(Part 6) (Both Treatment & Waitlist Control Groups) 1-month after completing the intervention the same battery as in Part 1 and Part 4 taking about 30 - 45 minutes will be completed.

(Waitlist control group) Upon completion of the 1-month follow-up assessment, the waitlist control group will be offered the opportunity to take part in the online intervention.

(Part 7) (Treatment Group only) 3-months after completing the intervention, a final Qualtrics link to complete the same battery as in Part 1, 4, and 6 taking about 30 - 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Chiari Malformation
* Access to the internet
* Be willing to commit approximately an hour a week for 8 weeks to engage in the intervention and homework
* Experience persistent pain for a minimum of 3-months
* Rate their pain intensity as greater than a 3 on a scale from 1-10
* Be stable on psychotropic medication for the past 3 months (if taking psychotropic medication)

Exclusion Criteria:

* Blindness
* Currently receiving Acceptance or Commitment Therapy or Cognitive Behavioral Therapy
* Have active suicidal ideations
* Diagnosed with a severe psychiatric disorder including bipolar disorder and schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in pain interference assessed by the Brief Pain Inventory Short-form over time | Assessed at baseline and weekly for 8-weeks, also assessed at the beginning of week 9, and 1-month and 3-months after the completion of the intervention
  This 9-item inventory assesses pain severity and pain interference over the past 24 hours. "Worst," "least," "average," and "current" pain severity are assessed. Pain interference items are measured on a scale from 0 - 10 (0 = Does not interfere, 10 = Completely interferes) and assesses the degree of pain interference in seven daily activities including general activity, walking, work, mood, enjoyment of life, relationships with others, and sleep. Prior research has demonstrated good internal validity and reliability in chronic pain samples.
Change in psychological flexibility assessed by the Acceptance and Action Questionnaire II over time | Assessed at baseline and weekly for 8-weeks, also assessed at the beginning of week 9, and 1-month and 3-months after the completion of the intervention
  This 7-item inventory is measured on a Likert scale (1 = never true, 7 = always true) and is the most commonly utilized measure of experiential avoidance and psychological flexibility. There is no specified time domain that this questionnaire evaluates. This measure assesses negative evaluations of emotions, avoidance of difficult thoughts and emotions, and behavioral modifications while in the context of challenging thoughts or feelings and has demonstrated good validity, and test re-test reliability
Change in sleep dysfunction assessed by the Insomnia Severity Index over time | Assessed at baseline and weekly for 8-weeks, also assessed at the beginning of week 9, and 1-month and 3-months after the completion of the intervention
  This 7-item index is used to capture perception of nocturnal and diurnal symptoms of insomnia over the past week. It specifically examines difficulties initiating sleep, maintaining sleep, and waking up too early, as well as satisfaction with current sleep, the perceived impact poor sleep has on quality of life and daily functioning, and distress related with sleep difficulties.
Change in sleep dysfunction assessed by the Daily Sleep Diary over time | Assessed for 7 days prior to the intervention and for 7 days following the intervention.
  This 12-question daily sleep diary assesses sleep duration, efficiency, and quality over the past night, these questions were used in a previous study (Tang, Goodchild, Sanborn, Howard, & Salkovskis, 2012). Questions include bedtime, rise time, how long it took to fall asleep, number of wake times (disrupted sleep maintenance), and length of time asleep. Additionally, a rating of quality of sleep (0 = very poor, 10 = very good), cognitive arousal (i.e., racing thoughts prior to bed), somatic arousal (i.e., feeling restless or jittery prior to bed), level of current pain (0 = no pain at all, 10 = a lot of pain), predicted amount of pain over the next day (0 = no pain at all, 10 = a lot of pain), and mood (0 = very bad mood, 10 = very good mood) is assessed.
Change in depression and anxiety assessed by the Depression Anxiety and Stress Scale-21 over time | Assessed at baseline and weekly for 8-weeks, also assessed at the beginning of week 9, and 1-month and 3-months after the completion of the intervention
  This 21-item measure that assesses depression, anxiety, and stress levels over the past week (Lovibond, Lovibond, & Australia, 1995). Internal consistencies for depression, anxiety, and stress in prior research has been good (Taylor, Lovibond, Nicholas, Cayley, & Wilson, 2005). In chronic pain samples the scale has demonstrated good internal consistency at the group level (Parkitny et al., 2012). Additionally, this measure does not include somatic symptoms in the depression scale, which prevents the depression score from being artificially inflated based on pain symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L Delahanty, PhD., Principal Investigator — Kent State University
Locations (1):
- Kent state University, Kent, Ohio, United States

REFERENCES:
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Buhrman M, Skoglund A, Husell J, Bergstrom K, Gordh T, Hursti T, Bendelin N, Furmark T, Andersson G. Guided internet-delivered acceptance and commitment therapy for chronic pain patients: a randomized controlled trial. Behav Res Ther. 2013 Jun;51(6):307-15. doi: 10.1016/j.brat.2013.02.010. Epub 2013 Mar 14. PMID 23548250
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carpenter JS, Andrykowski MA. Psychometric evaluation of the Pittsburgh Sleep Quality Index. J Psychosom Res. 1998 Jul;45(1):5-13. doi: 10.1016/s0022-3999(97)00298-5. PMID 9720850
- [Background] Cleeland, D. C. S. (2005). The Brief Pain Inventory- Short Form. 38.
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hayes S, Hogan M, Dowd H, Doherty E, O'Higgins S, Nic Gabhainn S, MacNeela P, Murphy AW, Kropmans T, O'Neill C, Newell J, McGuire BE. Comparing the clinical-effectiveness and cost-effectiveness of an internet-delivered Acceptance and Commitment Therapy (ACT) intervention with a waiting list control among adults with chronic pain: study protocol for a randomised controlled trial. BMJ Open. 2014 Jul 2;4(7):e005092. doi: 10.1136/bmjopen-2014-005092. PMID 24993763
- [Background] Kristjansdottir OB, Fors EA, Eide E, Finset A, Stensrud TL, van Dulmen S, Wigers SH, Eide H. A smartphone-based intervention with diaries and therapist-feedback to reduce catastrophizing and increase functioning in women with chronic widespread pain: randomized controlled trial. J Med Internet Res. 2013 Jan 7;15(1):e5. doi: 10.2196/jmir.2249. PMID 23291270
- [Background] Kroenke K, Wu J, Bair MJ, Krebs EE, Damush TM, Tu W. Reciprocal relationship between pain and depression: a 12-month longitudinal analysis in primary care. J Pain. 2011 Sep;12(9):964-73. doi: 10.1016/j.jpain.2011.03.003. Epub 2011 Jun 16. PMID 21680251
- [Background] Lin J, Klatt LI, McCracken LM, Baumeister H. Psychological flexibility mediates the effect of an online-based acceptance and commitment therapy for chronic pain: an investigation of change processes. Pain. 2018 Apr;159(4):663-672. doi: 10.1097/j.pain.0000000000001134. PMID 29320375
- [Background] Lovibond, S. H., Lovibond, P. F., & Australia, P. F. of. (1995). Manual for the depression anxiety stress scales. Retrieved from http://trove.nla.gov.au/version/46688692
- [Background] Parkitny L, McAuley JH, Walton D, Pena Costa LO, Refshauge KM, Wand BM, Di Pietro F, Moseley GL. Rasch analysis supports the use of the depression, anxiety, and stress scales to measure mood in groups but not in individuals with chronic low back pain. J Clin Epidemiol. 2012 Feb;65(2):189-98. doi: 10.1016/j.jclinepi.2011.05.010. Epub 2011 Sep 1. PMID 21889306
- [Background] Simister HD, Tkachuk GA, Shay BL, Vincent N, Pear JJ, Skrabek RQ. Randomized Controlled Trial of Online Acceptance and Commitment Therapy for Fibromyalgia. J Pain. 2018 Jul;19(7):741-753. doi: 10.1016/j.jpain.2018.02.004. Epub 2018 Mar 2. PMID 29481976
- [Background] Smith BW, Strahle J, Bapuraj JR, Muraszko KM, Garton HJ, Maher CO. Distribution of cerebellar tonsil position: implications for understanding Chiari malformation. J Neurosurg. 2013 Sep;119(3):812-9. doi: 10.3171/2013.5.JNS121825. Epub 2013 Jun 14. PMID 23767890
- [Background] Smith MT, Huang MI, Manber R. Cognitive behavior therapy for chronic insomnia occurring within the context of medical and psychiatric disorders. Clin Psychol Rev. 2005 Jul;25(5):559-92. doi: 10.1016/j.cpr.2005.04.004. PMID 15970367
- [Background] Tang NK, Goodchild CE, Sanborn AN, Howard J, Salkovskis PM. Deciphering the temporal link between pain and sleep in a heterogeneous chronic pain patient sample: a multilevel daily process study. Sleep. 2012 May 1;35(5):675-87A. doi: 10.5665/sleep.1830. PMID 22547894
- [Background] Taylor R, Lovibond PF, Nicholas MK, Cayley C, Wilson PH. The utility of somatic items in the assessment of depression in patients with chronic pain: a comparison of the Zung Self-Rating Depression Scale and the Depression Anxiety Stress Scales in chronic pain and clinical and community samples. Clin J Pain. 2005 Jan-Feb;21(1):91-100. doi: 10.1097/00002508-200501000-00011. PMID 15599136
- [Background] Trompetter HR, Bohlmeijer ET, Veehof MM, Schreurs KM. Internet-based guided self-help intervention for chronic pain based on Acceptance and Commitment Therapy: a randomized controlled trial. J Behav Med. 2015 Feb;38(1):66-80. doi: 10.1007/s10865-014-9579-0. Epub 2014 Jun 13. PMID 24923259
- [Background] van Hecke O, Torrance N, Smith BH. Chronic pain epidemiology and its clinical relevance. Br J Anaesth. 2013 Jul;111(1):13-8. doi: 10.1093/bja/aet123. PMID 23794640